CLINICAL TRIAL: NCT03369951
Title: A Phase IV Open-Label Pharmacokinetic Study of Minocycline for Injection Following a Single Infusion in Critically-Ill Adults (ACUMIN)
Brief Title: Minocycline Pharmacokinetics (ACUMIN)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16-0011; 2UM1AI104681-08 (NIH)
Record Dates: First submitted 2017-12-07; First posted 2017-12-12 (Actual); Results first posted 2020-08-27 (Actual); Last update posted 2020-12-03 (Actual); Status verified 2017-12-04

CONDITIONS: Bacterial Infection
Keywords: ACUMIN; Infusion; Injection; Minocycline; Pharmacokinetic; PK
MeSH Terms: conditions — Bacterial Infections; cyclopia sequence | interventions — Minocycline

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Minocin® IV (Experimental): 200 mg minocycline hydrochloride IV infusion over approximately 60 minutes, n=50
  Interventions: Drug: Minocycline

INTERVENTIONS:
Drug: Minocycline — Minocycline is a semisynthetic derivative of tetracycline and is indicated for the treatment of infections due to susceptible isolates of designated microorganisms.

SUMMARY:
This is a Phase IV, multi-center open-label pharmacokinetic trial studying the pharmacokinetics and pharmacodynamics of a single dose of Minocin IV. Up to 67 subjects will be enrolled to obtain 50 evaluable, ICU patients who are already receiving antimicrobial therapy for a known or suspected Gram-negative infection. The entire study duration will be approximately 16 months and each subject participation duration will be approximately 2 days. The study will be conducted at approximately 13 clinical sites. Each subject will receive a single 200 mg dose of Minocin IV infused over approximately 60 minutes. Each subject will have 7 PK samples collected (1 pre-dose, 6 post-dose) at designated time points over a ~48 hour period following the start of the Minocin IV infusion. The primary objectives are: 1) To characterize minocycline PK at the population level in critically-ill adults, with illness known or suspected to be caused by infection with Gram-negative bacteria and 2) To assess patient-level and clinical covariates associated with minocycline pharmacokinetic properties in critically-ill adults, with illness known or suspected to be caused by infection with Gram-negative bacteria.

DETAILED DESCRIPTION:
This is a Phase IV, multi-center open-label pharmacokinetic trial studying the pharmacokinetics and pharmacodynamics of a single dose of Minocin IV. Up to 67 subjects will be enrolled to obtain 50 evaluable, ICU patients who are already receiving antimicrobial therapy for a known or suspected Gram-negative infection. The entire study duration will be approximately 16 months and each subject participation duration will be approximately 2 days. The study will be conducted at approximately 13 clinical sites. Each subject will receive a single 200 mg dose of Minocin IV infused over approximately 60 minutes. Each subject will have 7 PK samples collected (1 pre-dose, 6 post-dose) at designated time points over a ~48 hour period following the start of the Minocin IV infusion. The primary objectives are: 1) To characterize minocycline PK at the population level in critically-ill adults, with illness known or suspected to be caused by infection with Gram-negative bacteria and 2) To assess patient-level and clinical covariates associated with minocycline pharmacokinetic properties in critically-ill adults, with illness known or suspected to be caused by infection with Gram-negative bacteria. Up to 67 subjects will be enrolled in order to obtain 50 PK evaluable subjects in the study. To be considered PK evaluable, a subject must receive the full infusion of study drug, and is required to have at least 3 PK samples collected in the first 12 hours post dose and at least 1 PK sample collected 24-48 hours post dose. Subjects who are dosed with minocycline but do not meet this PK sampling requirement will still be included in the population PK analysis, but an additional subject will be enrolled as a replacement to meet the goal of having 50 PK evaluable subjects with intensive PK sampling.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female > / = 18 years of age.
2. Subject is in the ICU, or is being admitted to the ICU.
3. Known or suspected Gram-negative infection for which the subject is receiving systemic antibiotics, and which was the reason for admission to the ICU, or reason for persistent need for ICU care.
4. Expectation, in the judgment of the investigator, that the subject will remain admitted in the hospital for at least 48 hours following enrollment and that all study procedures will be completed.
5. Expectation that intravenous access will be sufficient for drug infusion and either intravenous or arterial access will be sufficient to allow for all protocol required blood sampling to occur.
6. The subject, or legally authorized representative (LAR), is able and willing to provide signed informed consent.

Exclusion Criteria:

1. History of significant hypersensitivity or allergic reaction to tetracycline antibiotics.
2. Receipt of oral or intravenous tetracycline class drugs within 7 days of enrollment (e.g., minocycline, tetracycline, tigecycline, doxycycline).
3. Use of isotretinoin within 2 weeks of enrollment into the study.
4. Major surgery* within 48 hours prior to enrollment.

   *Major surgery is defined as "the opening of either a body cavity or the mesenchymal barrier, using general anesthesia".
5. Pregnant or breastfeeding women.
6. Patient is being treated for intracranial hypertension.
7. Any condition that, in the judgment of the investigator, precludes participation because it could affect subject safety.*

   *Subjects on, or who may be considered for Renal Replacement Therapy (RRT) during the study period are not excluded from participating in the study.
8. Receipt of an investigational study product within 7 days prior to enrollment. Investigator discretion should be used when longer acting agents have been used in the previous 30 days.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2018-03-28 (Actual); Primary Completion 2019-07-20 (Actual); Study Completion 2019-07-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (15):
- United States (15):
  - Emory Decatur Hospital - Clinical Trials - Immunology/Infectious Disease, Decatur, Georgia
  - Northwestern Memorial Hospital - ICU, Chicago, Illinois
  - Northwestern Medicine - Department of Obstetrics and Gynecology - Division of Female Pelvic Medicine and Reconstructive Surgery, Chicago, Illinois
  - University of Kentucky - UK Albert B Chandler Hospital, Lexington, Kentucky
  - University of Louisville School of Medicine - Surgery, Louisville, Kentucky
  - Henry Ford Health System - Henry Ford Hospital, Detroit, Michigan
  - William Beaumont Hospital - Royal Oak Campus - Infectious Disease, Royal Oak, Michigan
  - Washington University School of Medicine in St. Louis - Infectious Diseases, St Louis, Missouri
  - Duke University School of Medicine - Duke Clinical Research Institute - Duke Clinical Research Unit, Durham, North Carolina
  - Duke University Hospital - Duke Medicine Pavilion - MICU, Durham, North Carolina
  - East Carolina University - Infectious Diseases and Tropical/Travel Medicine Clinic, Greenville, North Carolina
  - University of Cincinnati College of Medicine - Division of Infectious Diseases, Cincinnati, Ohio
  - Case Western Reserve University School of Medicine - Medicine - Infectious Diseases and HIV Medicine, Cleveland, Ohio
  - Oregon Health and Science University - Division of Pulmonary and Critical Care Medicine, Portland, Oregon
  - University of Pittsburgh - Medicine - Infectious Diseases, Pittsburgh, Pennsylvania

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from those presenting at the ICU critically-ill with illness known or suspected to be caused by infection with Gram-negative bacteria. Enrollment occurred between 28MAR2018 and 18JUL2019.
Groups:
- Minocin® IV: 200 mg minocycline hydrochloride IV infusion over approximately 60 minutes
  Minocycline: Minocycline is a semisynthetic derivative of tetracycline and is indicated for the treatment of infections due to susceptible isolates of designated microorganisms.
Period: Overall Study
Arm/Group | Minocin® IV
Started | 58
Received Study Drug | 57
Completed | 52
Not Completed | 6
Not completed — Withdrawal by Subject | 3
Not completed — Death | 1
Not completed — Lost to Follow-up | 1
Not completed — Protocol Violation | 1

BASELINE CHARACTERISTICS:
Population: All subjects enrolled and receiving study product are included in the baseline analysis population description.
Arm/Group | Minocin® IV
Number analyzed (Participants) | 57
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 29
  >=65 years | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.6 (15.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25
  Male | 32
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 56
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 21
  White | 35
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 57
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 31.1 (10.46)

OUTCOME MEASURES:

1. Primary Outcome: Calculated Exposure Measures for Area Under the Curve 0 to 24 Hours After a Dose (AUC0-24)
Description: Total AUC0-24 is defined as area under the plasma minocycline concentration-time curve from 0 to 24 hours after a dose (milligrams x hours per liter (mg•hr/L)). Patient dosing histories along with the individual post-hoc PK parameters were used to generate total concentration-time profiles. The AUC0-24 was calculated using numerical integration using the data from 0 to 24 hours post-dose.
Time Frame: Pre-dose, immediately after infusion termination (~1 hour) and at 4, 12, and 24 hours post dose
Population: PK population which is defined as participants who (1) received the full infusion of study drug, (2) had at least one PK specimen was processed per the Manual of Procedures, and (3) had at least one such sample provided a quantifiable minocycline concentration available for analysis.
Measure: Mean (Standard Deviation); unit: mg·hr/L
Arm/Group | Minocin® IV
Number analyzed (Participants) | 55
mg·hr/L | 24.3 (7.88)

2. Primary Outcome: Calculated Exposure Measures for Area Under the Curve From 0 to Infinity (AUC0-inf) Using Free-drug Concentrations
Description: Free-drug (unbound) AUC0-inf is defined as area under the plasma minocycline concentration-time curve from 0 to infinity after a dose (mg•hr/L). Patient dosing histories along with the individual post-hoc PK parameters were used to generate unbound concentration-time profiles. The AUC0-inf was calculated as Dose/CL.
Time Frame: Pre-dose, immediately after infusion termination (~1 hour) and at 4, 12, 24, 36, and 48 post dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg·hr/L
Arm/Group | Minocin® IV
Number analyzed (Participants) | 55
mg·hr/L | 14.1 (6.68)

3. Primary Outcome: Calculated Exposure Measures for Area Under the Curve From 0 to Infinity (AUC0-inf) Using Total-drug Concentrations
Description: Total AUC0-inf is defined as area under the plasma minocycline concentration-time curve from 0 to infinity after a dose (mg•hr/L). Patient dosing histories along with the individual post-hoc PK parameters were used to generate total concentration-time profiles. The AUC0-inf was calculated as Dose/CL.
Time Frame: Pre-dose, immediately after infusion termination (~1 hour) and at 4, 12, 24, 36, and 48 post dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg·hr/L
Arm/Group | Minocin® IV
Number analyzed (Participants) | 55
mg·hr/L | 46.6 (19.7)

4. Primary Outcome: Calculated Exposure Measures for Area Under the Curve to the Last Quantifiable Sample (AUC0-last)
Description: AUC0-last is defined as the area under the plasma minocycline concentration-time curve from 0 to the time of the last quantifiable sample after a dose (mg•hr/L). This was not calculated for the primary outcome measure using the individual post-hoc PK parameters, however was calculated as part of the Non-compartmental analysis using the linear trapezoidal rule (linear up, log down calculation method).
Time Frame: Pre-dose, immediately after infusion termination (~1 hour) and at 4, 12, 24, 36, and 48 post dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg·h/L
Arm/Group | Minocin® IV
Number analyzed (Participants) | 51
mg·h/L | 10.5 (3.91)

5. Primary Outcome: Calculated Exposure Measures for Maximum Plasma Concentration (Cmax)
Description: Total-drug Cmax is defined as the maximum plasma total minocycline concentration (mg/L) Patient dosing histories along with the individual post-hoc PK parameters were used to generate total concentration-time profiles. Total Cmax was calculated for each simulated patient as the maximum simulated concentration.
Time Frame: Pre-dose, immediately after infusion termination (~1 hour) and at 4, 12, 24, 36, and 48 post dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Minocin® IV
Number analyzed (Participants) | 55
mg/L | 2.58 (1.33)

6. Primary Outcome: Calculated Exposure Measures for Plasma Concentration at 24 Hours After Dose (C24)
Description: Total-drug C24 is defined as total plasma minocycline concentration at 24 hours after a dose (mg/L). Patient dosing histories along with the individual post-hoc PK parameters were used to generate total concentration-time profiles. The total C24 were calculated for each simulated patient as the simulated concentration at 24 hours after dose.
Time Frame: Pre-dose, immediately after infusion termination (~1 hour) and at 4, 12, and 24 hours post dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Minocin® IV
Number analyzed (Participants) | 55
mg/L | 0.603 (0.225)

7. Primary Outcome: Individual Post-hoc PK Parameter Estimates for Area Under the Curve 0 to 24 Hours After a Dose (AUC0-24)
Description: Total AUC0-24 is defined as area under the plasma minocycline concentration-time curve from 0 to 24 hours after a dose (mg•hr/L). Patient dosing histories along with the individual post-hoc PK parameters were used to generate total concentration-time profiles. The AUC0-24 was calculated for each individual using numerical integration using the data from 0 to 24 hours post-dose. Summary statistics were calculated using the individual post-hoc parameters and reported as calculated exposure measures.
Time Frame: Pre-dose, immediately after infusion termination (~1 hour) and at 4, 12, and 24 hours post dose
Population: Individual post-hoc PK parameter estimate for AUC0-24 was calculated for each patient, summarized by mean and standard deviation, and reported as outcome measure 1 calculated exposure measures for area under the curve 0 to 24 hours after a dose (AUC0-24).
Arm/Group | Minocin® IV
Number analyzed (Participants) | 0

8. Primary Outcome: Individual Post-hoc PK Parameter Estimates for Area Under the Curve From 0 to Infinity (AUC0-inf) Using Free-drug Concentrations
Description: Free-drug (unbound) AUC0-inf is defined as area under the plasma minocycline concentration-time curve from 0 to infinity after a dose (mg•hr/L). Patient dosing histories along with the individual post-hoc PK parameters were used to generate unbound concentration-time profiles. The AUC0-inf was calculated for each individual as Dose/CL. Summary statistics were calculated using the individual post-hoc parameters and reported as calculated exposure measures.
Time Frame: Pre-dose, immediately after infusion termination (~1 hour) and at 4, 12, 24, 36, and 48 post dose
Population: Individual post-hoc PK parameter estimate for free-drug AUC0-inf was calculated for each patient, summarized by mean and standard deviation, and reported as outcome measure 2 Calculated exposure measures for area under the curve from 0 to infinity (AUC0-inf) using free-drug concentrations.
Arm/Group | Minocin® IV
Number analyzed (Participants) | 0

9. Primary Outcome: Individual Post-hoc PK Parameter Estimates for Area Under the Curve From 0 to Infinity (AUC0-inf) Using Total-drug Concentrations
Description: Total AUC0-inf is defined as area under the plasma minocycline concentration-time curve from 0 to infinity after a dose (mg•hr/L). Patient dosing histories along with the individual post-hoc PK parameters were used to generate total concentration-time profiles. The AUC0-inf was calculated for each individual as Dose/CL. Summary statistics were calculated using the individual post-hoc parameters and reported as calculated exposure measures.
Time Frame: Pre-dose, immediately after infusion termination (~1 hour) and at 4, 12, 24, 36, and 48 post dose
Population: Individual post-hoc PK parameter estimate for total AUC0-inf was calculated for each patient, summarized by mean and standard deviation, and reported as outcome measure 3 calculated exposure measures for area under the curve from 0 to infinity (AUC0-inf) using total-drug concentrations.
Arm/Group | Minocin® IV
Number analyzed (Participants) | 0

10. Primary Outcome: Individual Post-hoc PK Parameter Estimates for Area Under the Curve to the Last Quantifiable Sample (AUC0-last)
Description: AUC0-last is defined as the area under the plasma minocycline concentration-time curve from 0 to the time of the last quantifiable sample after a dose (mg•hr/L). This was not calculated of the primary outcome measure for the population PK model, however was calculated as part of the Non-compartmental analysis using the linear trapezoidal rule (linear up, log down calculation method).
Time Frame: Pre-dose, immediately after infusion termination (~1 hour) and at 4, 12, 24, 36, and 48 post dose
Population: Individual AUC0-last were calculated as part of the Non-compartmental analysis using the linear trapezoidal rule, summarized by mean and standard deviation, and reported as outcome measure 4 calculated exposure measures for area under the curve to the last quantifiable sample (AUC0-last).
Arm/Group | Minocin® IV
Number analyzed (Participants) | 0

11. Primary Outcome: Individual Post-hoc PK Parameter Estimates for Maximum Plasma Concentration (Cmax)
Description: Total-drug Cmax is defined as the maximum plasma total minocycline concentration (mg/L). Patient dosing histories along with the individual post-hoc PK parameters were used to generate total concentration-time profiles. The Individual post-hoc PK parameter estimate for total Cmax was calculated for each simulated patient as the maximum simulated concentration. Summary statistics were calculated using the individual post-hoc parameters and reported as calculated exposure measures.
Time Frame: Pre-dose, immediately after infusion termination (~1 hour) and at 4, 12, 24, 36, and 48 post dose
Population: Individual post-hoc PK parameter estimate for total-drug Cmax was calculated for each patient, summarized by mean and standard deviation, and reported as outcome measure 5 calculated exposure measures for maximum plasma concentration (Cmax).
Arm/Group | Minocin® IV
Number analyzed (Participants) | 0

12. Primary Outcome: Individual Post-hoc PK Parameter Estimates for Plasma Concentration at 24 Hours After Dose (C24)
Description: Total-drug C24 is defined as total Plasma minocycline concentration at 24 hours after a dose (mg/L). Patient dosing histories along with the individual post-hoc PK parameters were used to generate total concentration-time profiles. The Individual post-hoc PK parameter estimates for the total C24 were calculated for each simulated patient as the simulated concentration at 24 hours after dose. Summary statistics were calculated using the individual post-hoc parameters and reported as calculated exposure measures.
Time Frame: Pre-dose, immediately after infusion termination (~1 hour) and at 4, 12, and 24 hours post dose
Population: Individual post-hoc PK parameter estimate for total-drug C24 was calculated for each patient, summarized by mean and standard deviation, and reported as outcome measure 6 calculated exposure measures for plasma concentration at 24 hours after dose (C24).
Arm/Group | Minocin® IV
Number analyzed (Participants) | 0

13. Primary Outcome: Magnitude of the Inter-individual Variability for Central Volume of Distribution (Vc)
Description: Vc was estimated from the structural two-compartment population PK model with constant fraction unbound (fub) which was used to characterize the total and unbound minocycline concentration-time data from ICU patients. The model was developed on using nonlinear mixed effects modeling on PK time points collected up to 48 hours after a single-dose on Day 1. Magnitude of the inter-individual variability is expressed as percent coefficient of variation (%CV).
Time Frame: Pre-dose, immediately after infusion termination (~1 hour) and at 4, 12, 24, 36, and 48 post dose
Population: as for outcome 1
Measure: Number; unit: %CV
Arm/Group | Minocin® IV
Number analyzed (Participants) | 55
%CV | 49.9

14. Primary Outcome: Magnitude of the Inter-individual Variability for Distribution Clearance (CLd)
Description: CLd was estimated from the structural two-compartment population PK model with constant fraction unbound (fub) which was used to characterize the total and unbound minocycline concentration-time data from ICU patients. The model was developed on using nonlinear mixed effects modeling on PK time points collected up to 48 hours after a single-dose on Day 1. The standard error of the mean as fixed. Magnitude of the inter-individual variability is expressed as percent coefficient of variation (CV%).
Time Frame: Pre-dose, immediately after infusion termination (~1 hour) and at 4, 12, 24, 36, and 48 post dose
Population: as for outcome 1
Measure: Number; unit: %CV
Arm/Group | Minocin® IV
Number analyzed (Participants) | 55
%CV | 0

15. Primary Outcome: Magnitude of the Inter-individual Variability for Free-drug Clearance (CL)
Description: Unbound minocycline concentration is determined as the product of total minocycline concentrations and fub. Total minocycline concentrations and fub were estimated from the structural two-compartment population PK model with constant fraction unbound (fub) which was used to characterize the total and unbound minocycline concentration-time data from ICU patients. Magnitude of the inter-individual variability is expressed as percent coefficient of variation (%CV).
Time Frame: Pre-dose, immediately after infusion termination (~1 hour) and at 4, 12, 24, 36, and 48 post dose
Population: The model was fit with total drug clearance and then fraction unbound so the magnitude of the inter-individual variability was estimated for those parameters rather than free-drug.
Arm/Group | Minocin® IV
Number analyzed (Participants) | 0

16. Primary Outcome: Magnitude of the Inter-individual Variability for Peripheral Volume of Distribution (Vp)
Description: Vp was estimated from the structural two-compartment population PK model with constant fraction unbound (fub), which was used to characterize the total and unbound minocycline concentration-time data from ICU patients. The model was developed on using nonlinear mixed effects modeling on PK time points collected up to 48 hours after a single-dose on Day 1.
Time Frame: Pre-dose, immediately after infusion termination (~1 hour) and at 4, 12, 24, 36, and 48 post dose
Population: as for outcome 1
Measure: Number; unit: %CV
Arm/Group | Minocin® IV
Number analyzed (Participants) | 55
%CV | 34.2

17. Primary Outcome: Magnitude of the Inter-individual Variability for Total-drug Clearance (CL)
Description: CL was estimated from the structural two-compartment population PK model with constant fraction unbound (fub) which was used to characterize the total and unbound minocycline concentration-time data from ICU patients. The model was developed on using nonlinear mixed effects modeling on PK time points collected up to 48 hours after a single-dose on Day 1. Magnitude of the inter-individual variability is expressed as percent coefficient of variation (%CV).
Time Frame: Pre-dose, immediately after infusion termination (~1 hour) and at 4, 12, 24, 36, and 48 post dose
Population: as for outcome 1
Measure: Number; unit: %CV
Arm/Group | Minocin® IV
Number analyzed (Participants) | 55
%CV | 45.6

18. Primary Outcome: Population Mean PK Parameter Estimates for Central Volume of Distribution (Vc)
Description: Vc was estimated from the structural two-compartment population PK model with constant fraction unbound (fub) which was used to characterize the total and unbound minocycline concentration-time data from ICU patients. The model was developed on using nonlinear mixed effects modeling on PK time points collected up to 48 hours after a single-dose on Day 1.
Time Frame: Pre-dose, immediately after infusion termination (~1 hour) and at 4, 12, 24, 36, and 48 post dose
Population: as for outcome 1
Measure: Mean (Standard Error); unit: L
Arm/Group | Minocin® IV
Number analyzed (Participants) | 55
L | 74.5 (6.60)

19. Primary Outcome: Population Mean PK Parameter Estimates for Distribution Clearance (CLd)
Description: CLd was estimated from the structural two-compartment population PK model with constant fraction unbound (fub), which was used to characterize the total and unbound minocycline concentration-time data from ICU patients. The model was developed on using nonlinear mixed effects modeling on PK time points collected up to 48 hours after a single-dose on Day 1.
Time Frame: Pre-dose, immediately after infusion termination (~1 hour) and at 4, 12, 24, 36, and 48 post dose
Population: as for outcome 1
Measure: Mean (Standard Error); unit: L/hr
Arm/Group | Minocin® IV
Number analyzed (Participants) | 55
L/hr | 16.0 (8.66)

20. Primary Outcome: Population Mean PK Parameter Estimates for Free-drug Clearance (CL)
Description: Unbound minocycline concentration is determined as the product of total minocycline concentrations and fub. Total minocycline concentrations and fub were estimated from the structural two-compartment population PK model with constant fraction unbound (fub) which was used to characterize the total and unbound minocycline concentration-time data from ICU patients.
Time Frame: Pre-dose, immediately after infusion termination (~1 hour) and at 4, 12, 24, 36, and 48 post dose
Population: as for outcome 1
Measure: Mean (Standard Error); unit: L/hr
Arm/Group | Minocin® IV
Number analyzed (Participants) | 55
L/hr | 1.32 (0)

21. Primary Outcome: Population Mean PK Parameter Estimates for Peripheral Volume of Distribution (Vp)
Description: as for outcome 16
Time Frame: Pre-dose, immediately after infusion termination (~1 hour) and at 4, 12, 24, 36, and 48 post dose
Population: as for outcome 1
Measure: Mean (Standard Error); unit: L
Arm/Group | Minocin® IV
Number analyzed (Participants) | 55
L | 58.9 (5.89)

22. Primary Outcome: Population Mean PK Parameter Estimates for Total-drug Clearance (CL)
Description: Total-drug clearance (CL) was estimated from the structural two-compartment population PK model with constant fraction unbound (fub), which was used to characterize the total and unbound minocycline concentration-time data from ICU patients. The model was developed on using nonlinear mixed effects modeling on PK time points collected up to 48 hours after a single-dose on Day 1.
Time Frame: Pre-dose, immediately after infusion termination (~1 hour) and at 4, 12, 24, 36, and 48 post dose
Population: as for outcome 1
Measure: Mean (Standard Error); unit: L/hr
Arm/Group | Minocin® IV
Number analyzed (Participants) | 55
L/hr | 4.7 (6.24)

ADVERSE EVENTS:
Time Frame: Serious Adverse Events (SAEs) were recorded and reported from the start of the Minocin IV infusion until 24 hours from the start of infusion.
Description: As this is an approved product at an approved dose, and the study is being performed in subjects in the ICU who were anticipated to have multiple events due to their underlying disease, only SAEs were captured in this protocol.
Arm/Group | Minocin® IV
All-Cause Mortality (participants affected / at risk) | 1/57
Serious Adverse Events (participants affected / at risk) | 1/57
Other Adverse Events (participants affected / at risk) | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Minocin® IV (N=57)
Cardio-Respiratory Arrest (Cardiac disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (3):
  • Study Protocol (2018-11-19): https://cdn.clinicaltrials.gov/large-docs/51/NCT03369951/Prot_000.pdf
  • Statistical Analysis Plan (2019-07-11): https://cdn.clinicaltrials.gov/large-docs/51/NCT03369951/SAP_001.pdf
  • Informed Consent Form (2019-06-03): https://cdn.clinicaltrials.gov/large-docs/51/NCT03369951/ICF_002.pdf